CLINICAL TRIAL: NCT03056885
Title: Does a Protective One Lung Ventilation Strategy Reduce the Inflammatory Cytokine Local Response After Pulmonary Resection?
Brief Title: Inflammatory Local Response During OLV: Protective vs Conventional Ventilation Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Mohsen Ibrahim, Medical Director, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3722/2015
Record Dates: First submitted 2017-02-12; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Ventilator-Induced Lung Injury; Inflammatory Response; Respiratory Complication
Keywords: one-lung ventilation; broncho-alveolar lavage; protective ventilation; cytokines; thoracic surgery
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional One-lung ventilation (Experimental): The patients received a Tidal volume of 10 ml/kg (based on Predicted body weight)
  Interventions: Other: Conventional One-Lung Ventilation
- Protective One-Lung Ventilation (Experimental): The patients received a Tidal volume of 5 ml/kg (based on Predicted body weight)
  Interventions: Other: Protective One-lung ventilation

INTERVENTIONS:
Other: Conventional One-Lung Ventilation — Vt 10 ml/kg
  Arms: Conventional One-lung ventilation
Other: Protective One-lung ventilation — Vt 5 ml/kg
  Arms: Protective One-Lung Ventilation

SUMMARY:
This study evaluates the local cytokine inflammatory response during one lung ventilation in patients undergoing pulmonary lobectomy or wedge resection. We compare two different ventilation strategies: a conventional strategy with a protective strategy.

DETAILED DESCRIPTION:
One-lung ventilation (OLV) is a ventilation procedure used for pulmonary resection often causing lung injury. International guidelines have recommended for years the use of conventional ventilation (CV) with high tidal volume (VT) (8-10 ml\kg).A body of recent evidences have shown that conventional ventilation can reduce systemic oxygenation, increase inflammatory products and cause lung tissue damage. In this study we compare the conventional strategy , consisted of Vt 10 mL/kg, with the protective strategy, consisted of Vt 5 mL/kg. Both Vt were based on predicted body weight (PBW). Broncho-alveolar lavages (BAL) are selectively performed in the dependent (ventilated) lung before and at the end of the OLV. The levels of pro-inflammatory (IL-1α, IL-1β, IL-6, IL-8, TNF) and anti-inflammatory (IL-2, IL-4, IL-10, INFγ) cytokines are evaluated. We also evaluate patients clinical outcomes in terms of incidence of postoperative respiratory complications and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective lobectomy and wedge resection

Exclusion Criteria:

* emergency surgery, pregnancy, patient refusal, inability to give consent, age ≤ 18 years and ≥ ASA IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2015-11-25 (Actual); Study Completion 2016-01-15 (Actual)

PRIMARY OUTCOMES:
local cytokine inflammatory response in the two study groups | Change from Baseline cytokines level and the end of surgery (about 60 minutes)
  The levels of cytokines were evaluated in broncho-alveolar lavage (BAL)

SECONDARY OUTCOMES:
incidence of postoperative respiratory in the two study groups | within 48 hours of the operation
  PaO2 /FIO 2 <300 mm Hg and /or the presence of newly developed lung lesions (lung infi ltration and atelectasis)
lenght of stay in the two study groups | 1 month
  lenght of hospital stay expressed in days

IPD SHARING:
Plan to Share IPD: No